CLINICAL TRIAL: NCT02201680
Title: Anxiety Level of Child and Parents During Preoperative Anesthesia Evaluation
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Prof. Dr. A. Pervin SUTAS BOZKURT, Prof. Dr., Istanbul University
Other Study IDs: 15112005; 31130 (Other: Cerrahpasa Medical Faculty Clinical Trials Ethics Committee)
Record Dates: First submitted 2014-07-12; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Anxiety State; Parent; Child
Keywords: anxiety; preoperative
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- parents and children: Anxiety tests

SUMMARY:
1. Appreciation of preoperative anxiety in children is important for the anesthesiologist.
2. Several factors defined to effect the anxiety levels preoperatively in children such as , age, previous medical encounters , education level and parental anxiety. 3. This information was tested for Turkish children during the preoperative anesthetic evaluation.

DETAILED DESCRIPTION:
1. Before the planned surgery all children accompanying parents filled a questionnaire about the demographics, marital status, economical conditions, education level and other diseases and operations in the family.
2. Both the parent and child filled State and Trait Anxiety tests specially prepared for adults Spielberger Anxiety tests and children defined and validation tests had already been proven.

Statistical analysis performed for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Legible

Exclusion Criteria:

* Illegible due to lack of education or eye diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children planned to undergo surgical procedures or diagnostic procedures under general anesthesia
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
children state anxiety | 1 hour
  Anxiety scores were filled within 1 hour no further evalution was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Rovnat Babazade, M.D., Principal Investigator — Istanbul University Cerrahpaşa Medical Faculty; Levent Kayaalp, Prof. Dr., Principal Investigator — Private Practice; Gurcan Gungor, M.D., Principal Investigator — Istanbul University; Burak Dogangun, Asoc. Prof, Principal Investigator — Istanbul University